CLINICAL TRIAL: NCT02511470
Title: The Use of an Audible Metronome Improves Chest Compression During Cardiopulmonary Resuscitation on a Pediatric Simulation Manikin
Brief Title: Use of a Metronome in Cardiopulmonary Resuscitation: A Simulation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nicklaus Children's Hospital f/k/a Miami Children's Hospital (Other)
Collaborators: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 1-806360-1
Record Dates: First submitted 2015-07-22; First posted 2015-07-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Cardiac Arrest
Keywords: Cardiopulmonary Resuscitation; Pediatric simulation study; Metronome
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPR with metronome on (Other): Participants will perform two minutes of uninterrupted chest compressions on a pediatric manikin with the metronome on. Data for compression rate and depth will be collected during this time interval.
  Interventions: Other: Metronome on
- CPR with metronome off (Other): Participants will perform two minutes of uninterrupted chest compressions on a pediatric manikin with the metronome off. Data for compression rate and depth will be collected during this time interval.
  Interventions: Other: Metronome off

INTERVENTIONS:
Other: Metronome on — Metronome on during participants performance of CPR on a pediatric manikin
  Arms: CPR with metronome on
Other: Metronome off — Metronome off during participants performance of CPR on a pediatric manikin
  Arms: CPR with metronome off

SUMMARY:
The purpose of this study is to determine if the use of a metronome improves chest compression rate and depth during cardiopulmonary resuscitation (CPR) on a pediatric manikin.

DETAILED DESCRIPTION:
The study will be conducted in the simulation laboratory at Miami Children's Hospital. Chest compressions will be performed on a compression pediatric simulator. It will consist of two main groups randomly assigned to chest compressions without an audible metronome and chest compressions with audible metronomic tones that beep 100 times per minute for chest compressions. The metronome will be used to coach the correct rate. The same people will complete both arms of the study at one visit. Specifically, the participants will do 2 minutes of chest compressions followed by a 15-minute break then another 2 minutes of chest compressions (to avoid fatigue) with an acceptable range for rate 90-110 BPM and depth of 38-51mm. The subjects will be informed about the metronome, but will not be informed about the measured variables, such as rate and depth of chest compressions. However, the participants will be reminded at the beginning of their visit about the PALS card, i.e. appropriate rate and depth. The use of "talking people noise" from YouTube will be played in the background to fully model a cardiac arrest scenario (to see if participants ignore the metronome) and will be used during each group session. A noise dosimeter will be used to ensure this noise level is the same for each scenario. The manikin's airway will be secured with an endotracheal tube with continuous ventilations so chest compressions can be continued without interruption. Recommendations for chest compression rate and depth are per Pediatric Advanced Life Support (PALS) according to the 2010 American Heart Association (AHA) guidelines.

Data will be collected via the manikin which will wirelessly transmit the data (chest compression rate and depth) to a computer. The manikin has CPR sensing and recording technology software built in. This software records sternum movement depth and rate of chest compressions. Criteria for adequate CPR quality are defined as compression rate between 90-110 per minute and compression depth between 38-51mm.

ELIGIBILITY:
Inclusion criteria:

* health professionals with a minimum of basic life support training according to the 2010 AHA guidelines capable of performing chest compressions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Metronome effect on compression rate and depth | Adequacy of chest compressions (in terms of rate and depth) under each intervention (with and without metronome) was assessed during two minutes
  The mean of the percentage of compressions that were within an adequate rate (90-110 per minute) and adequate depth (38-51mm) with and without the metronome.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Linares, MD, Principal Investigator — Nicklaus Children's Hospital f/k/a Miami Children's Hospital

REFERENCES:
- [Background] Abella BS, Sandbo N, Vassilatos P, Alvarado JP, O'Hearn N, Wigder HN, Hoffman P, Tynus K, Vanden Hoek TL, Becker LB. Chest compression rates during cardiopulmonary resuscitation are suboptimal: a prospective study during in-hospital cardiac arrest. Circulation. 2005 Feb 1;111(4):428-34. doi: 10.1161/01.CIR.0000153811.84257.59. PMID 15687130
- [Background] Al-Shamsi M, Al-Qurashi W, de Caen A, Bhanji F. Pediatric basic and advanced life support: an update on practice and education. Oman Med J. 2012 Nov;27(6):450-4. doi: 10.5001/omj.2012.108. PMID 23226814
- [Background] Bohn A, Weber TP, Wecker S, Harding U, Osada N, Van Aken H, Lukas RP. The addition of voice prompts to audiovisual feedback and debriefing does not modify CPR quality or outcomes in out of hospital cardiac arrest--a prospective, randomized trial. Resuscitation. 2011 Mar;82(3):257-62. doi: 10.1016/j.resuscitation.2010.11.006. Epub 2010 Dec 13. PMID 21146279
- [Background] Dine CJ, Gersh RE, Leary M, Riegel BJ, Bellini LM, Abella BS. Improving cardiopulmonary resuscitation quality and resuscitation training by combining audiovisual feedback and debriefing. Crit Care Med. 2008 Oct;36(10):2817-22. doi: 10.1097/CCM.0b013e318186fe37. PMID 18766092
- [Background] Fitzgerald KR, Babbs CF, Frissora HA, Davis RW, Silver DI. Cardiac output during cardiopulmonary resuscitation at various compression rates and durations. Am J Physiol. 1981 Sep;241(3):H442-8. doi: 10.1152/ajpheart.1981.241.3.H442. PMID 7282953
- [Background] Handley AJ, Handley SA. Improving CPR performance using an audible feedback system suitable for incorporation into an automated external defibrillator. Resuscitation. 2003 Apr;57(1):57-62. doi: 10.1016/s0300-9572(02)00400-8. PMID 12668300
- [Background] Hurst VW 4th, Whittam SW, Austin PN, Branson RD, Beck G. Cardiopulmonary resuscitation during spaceflight: examining the role of timing devices. Aviat Space Environ Med. 2011 Aug;82(8):810-3. doi: 10.3357/asem.2284.2011. PMID 21853860
- [Background] Jantti H, Silfvast T, Turpeinen A, Kiviniemi V, Uusaro A. Influence of chest compression rate guidance on the quality of cardiopulmonary resuscitation performed on manikins. Resuscitation. 2009 Apr;80(4):453-7. doi: 10.1016/j.resuscitation.2009.01.001. Epub 2009 Feb 8. PMID 19203821
- [Background] Kern KB, Hilwig RW, Berg RA, Ewy GA. Efficacy of chest compression-only BLS CPR in the presence of an occluded airway. Resuscitation. 1998 Dec;39(3):179-88. doi: 10.1016/s0300-9572(98)00141-5. PMID 10078808
- [Background] Kern KB. Cardiopulmonary resuscitation without ventilation. Crit Care Med. 2000 Nov;28(11 Suppl):N186-9. doi: 10.1097/00003246-200011001-00003. PMID 11098942
- [Background] Kern KB, Stickney RE, Gallison L, Smith RE. Metronome improves compression and ventilation rates during CPR on a manikin in a randomized trial. Resuscitation. 2010 Feb;81(2):206-10. doi: 10.1016/j.resuscitation.2009.10.015. Epub 2009 Nov 18. PMID 19926194
- [Background] Kleinman ME, Chameides L, Schexnayder SM, Samson RA, Hazinski MF, Atkins DL, Berg MD, de Caen AR, Fink EL, Freid EB, Hickey RW, Marino BS, Nadkarni VM, Proctor LT, Qureshi FA, Sartorelli K, Topjian A, van der Jagt EW, Zaritsky AL. Part 14: pediatric advanced life support: 2010 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2010 Nov 2;122(18 Suppl 3):S876-908. doi: 10.1161/CIRCULATIONAHA.110.971101. No abstract available. PMID 20956230
- [Background] Kramer-Johansen J, Myklebust H, Wik L, Fellows B, Svensson L, Sorebo H, Steen PA. Quality of out-of-hospital cardiopulmonary resuscitation with real time automated feedback: a prospective interventional study. Resuscitation. 2006 Dec;71(3):283-92. doi: 10.1016/j.resuscitation.2006.05.011. Epub 2006 Oct 27. PMID 17070980
- [Background] Matos RI, Watson RS, Nadkarni VM, Huang HH, Berg RA, Meaney PA, Carroll CL, Berens RJ, Praestgaard A, Weissfeld L, Spinella PC; American Heart Association's Get With The Guidelines-Resuscitation (Formerly the National Registry of Cardiopulmonary Resuscitation) Investigators. Duration of cardiopulmonary resuscitation and illness category impact survival and neurologic outcomes for in-hospital pediatric cardiac arrests. Circulation. 2013 Jan 29;127(4):442-51. doi: 10.1161/CIRCULATIONAHA.112.125625. Epub 2013 Jan 22. PMID 23339874
- [Background] Milander MM, Hiscok PS, Sanders AB, Kern KB, Berg RA, Ewy GA. Chest compression and ventilation rates during cardiopulmonary resuscitation: the effects of audible tone guidance. Acad Emerg Med. 1995 Aug;2(8):708-13. doi: 10.1111/j.1553-2712.1995.tb03622.x. PMID 7584749
- [Background] Ochoa FJ, Ramalle-Gomara E, Lisa V, Saralegui I. The effect of rescuer fatigue on the quality of chest compressions. Resuscitation. 1998 Jun;37(3):149-52. doi: 10.1016/s0300-9572(98)00057-4. PMID 9715774
- [Background] Young KD, Gausche-Hill M, McClung CD, Lewis RJ. A prospective, population-based study of the epidemiology and outcome of out-of-hospital pediatric cardiopulmonary arrest. Pediatrics. 2004 Jul;114(1):157-64. doi: 10.1542/peds.114.1.157. PMID 15231922
- [Derived] Zimmerman E, Cohen N, Maniaci V, Pena B, Lozano JM, Linares M. Use of a Metronome in Cardiopulmonary Resuscitation: A Simulation Study. Pediatrics. 2015 Nov;136(5):905-11. doi: 10.1542/peds.2015-1858. Epub 2015 Oct 12. PMID 26459645